CLINICAL TRIAL: NCT00190073
Title: Cutaneous Denervation in Alcoholic Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Other Study IDs: FEMH-94003; FEMH-94003
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Alcohol Abuse; Peripheral Neuropathy
Keywords: Epidermal nerves;protein gene product 9.5; ethanol
MeSH Terms: conditions — Alcoholism; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Peripheral neuropathy is a frequent neurological complication of chronic alcoholism. Most studies evaluated large-fiber involvement by nerve conduction studies (NCS). Since previous studies document the predominant injury of small myelinated and unmyelinated fibers in patients with alcoholic neuropathy, it will be imperative to know their prevalence and clinical significance. Moreover, the pathogenesis of alcoholic neuropathy, especially the roles of ethanol and its metabolites and thiamine, remains elusive. This proposal will be designed to understand the extent and clinical significance of cutaneous nerve degeneration in the skin of alcoholic patients and to investigate its pathogenesis. We will investigate cutaneous innervation by 3 mm punch skin biopsies with immunohistochemistry for protein gene product 9.5 and quantifying epidermal nerve density (END) in alcoholic patients. Patients will undergo clinical evaluation, quantitative sensory testing (QST), nerve conduction studies (NCS), and tests of sympathetic skin response (SSR) and beat-to-beat RR interval variability (RRIV). The prevalence of peripheral neuropathy in chronic alcoholic patients with emphasis on small-fiber involvement will be first evaluated. The sensitivity of punch skin biopsy, QST, SSR and RRIV tests, and NCS will be compared, and the correlations between END and psychophysic and electrodiagnostic parameters will be discussed. Subsequently, we will elucidate the clinical significance of END reduction in alcoholic patients. Patients with evidences of involvement of central nervous system will be excluded, and END will be correlated with clinical manifestations and neurological deficits. Finally, the role of ethanol and thiamine in alcoholic neuropathy will be further studied. To clarify the role of thiamine in alcoholic neuropathy, we will examine whether it has influences on small-fiber degeneration. This may provide important information in understanding the pathogenesis and designing optimal treatment for alcoholic neuropathy.

DETAILED DESCRIPTION:
Alcoholic patients and control subjects. Alcoholic patients will be recruited from neurologic clinics and ward at the Far Eastern Memorial Hospital, Taipei, Taiwan. A detailed clinical history that includes daily alcohol consumption, daily dietary intake, lifestyle, and occupation will be obtained from patients as well as their families. The inclusion criteria include daily uptake of at least 100 g ethanol for more than 3 years prior to the onset of neuropathic symptoms (Behse and Buchthal, 1977). All patients will undergo clinical and neurologic assessment, cranial MRI or CT, and neuropsychological evaluation to rule out CNS disorders, which interfere the evaluation of neuropathic symptoms and signs and psychophysic test. Laboratory investigations will include complete blood count, fasting plasma glucose, hemoglobin A1C, liver and renal function tests, ethanol level, tumor markers, antinuclear antibodies, complement factors, serum protein electrophoresis, thyroid function, human immunodeficiency virus, hepatitis virus, and vitamin B12 level. Thiamine status will be assessed at the time of the first referral to the hospital by measuring total thiamine concentration in whole blood by high performance liquid chromatography, as described elsewhere (Koike et al., 2001 and 2003). None of the patients will administrate thiamine at the time of determination. Age- and gender-matched control subjects will be retrieved from our database, who will be evaluated by detailed questionnaires and neurological examinations to exclude any neurological disorder or clinical neuropathy (McCarthy et al., 1995).

Skin biopsy. Skin biopsy will be performed following established procedures after informed consent has been obtained (McCarthy et al., 1995; Pan et al., 2003; Shun et al., 2004). Under local anesthesia with 2% lidocaine, punches 3mm in diameter will be taken from the following locations: (1) the extensor side of the distal forearm, 5 cm above the middle point of a line connecting the radial styloid process and the ulnar styloid process; and (2) the lateral side of the distal leg, 10 cm above the lateral malleolus. No suturing will be required, and the wounds will be covered with a piece of gauze. Wound healing takes 7-10 days, the same as would a typical abrasion wound. The protocol is under review by the Ethics Committee of Far Eastern Memorial Hospital.

Immunohistochemistry. For immunohistochemistry on freezing microtome sections, the skin samples will be fixed with 4% paraformaldehyde in 0.1M phosphate-buffered saline (PBS), pH 7.4, for 48 h (McCarthy et al., 1995; Hsieh et al., 2000). Sections of 50 mm perpendicular to the dermis will be cut on a sliding microtome (model 440E; Microm, Walldorf, Germany). They will be quenched with 1% H2O2, blocked with 5% normal goat serum, and incubated with rabbit antiserum to PGP 9.5 (UltraClone, UK, diluted 1: 1000 in 1% normal serum/Tris) at 4C for 16-24 h. After rinsing in Tris, sections will be incubated with biotinylated goat anti-rabbit IgG at room temperature for 1 h, followed by incubation with avidin-biotin complex (Vector, Burlingame, CA) for another hour. The reaction product will be demonstrated with chromogen SG (Vector, Burlingame, CA), and counterstained with eosin (Sigma, St. Louis, MO).

Quantitation of epidermal innervation. Epidermal innervation will be quantified following established protocols, and slides will be coded to ensure that measurements are blinded (Hsieh et al., 2000; Pan et al., 2003; Shun et al., 2004). PGP 9.5-immunoreactive nerve fibers in the epidermis of each section will be counted at a magnification of  40 with an Olympus BX40 microscope (Tokyo, Japan) through the depth of the entire section. Each individual nerve with branching points inside the epidermis will be counted as one. For epidermal nerves with branching points in the dermis, each individual nerve will be counted separately. The length of the epidermis along the upper margin of the stratum corneum in each section will be measured using Image-Pro PLUS (Media Cybernetics, Silver Spring, MD). END will therefore be derived and expressed as fibers/mm. For each tissue, there will be 48-50 sections, and all sections will be sequentially labeled. Every fifth section will be immunostained and quantified. The mean of values from these sections will be considered the END of the tissue specimen. In the distal leg, normative values from our laboratory (mean  SD, 5th percentile) of END are 11.16  3.70, 5.88 fibres/mm for subjects aged < 60 years and 7.64  3.08, 2.50 fibres/mm for subjects aged  60 years. The cut-off point of END is 5.88 and 2.50 fibres/mm in the two age groups, respectively.

Quantitative sensory testing. We will perform quantitative sensory testing (QST) with a Thermal Sensory Analyzer and Vibratory Sensory Analyzer (Medoc Advanced Medical System, Minneapolis, MN) to measure thresholds of warm, cold, and vibratory sensations following the established protocol (Pan et al., 2001; Pan et al., 2003; Yarnitsky and Ochoa, 1991). Briefly, the machine will deliver a stimulus of constant intensity which had been determined by the test algorithm. The intensity of the next stimulus will be either increased or decreased by a fixed ratio according to the response of the subject, i.e., whether or not the subject perceives the stimulus. Such procedures will be repeated until a pre-determined difference of intensity is reached. The mean intensity of the last two stimuli will be the threshold for the level method. Thermal thresholds recorded on the toe will be expressed as warm threshold temperature and cold threshold temperature, respectively. These temperatures will be compared with normative values (Pan et al., 2003). Vibratory thresholds recorded on the malleolus will be measured with similar algorithms. Normative values are documented previously and are similar to those of previous reports (Pan et al., 2001; Pan et al., 2003). Threshold values greater than the 95th percentile value for each age group will be considered abnormal.

Nerve conduction studies. NCS will be carried out in all patients with a Keypoint electromyographer following standardized methods (Pan et al., 2003). Amplitudes of compound muscle action potential (CMAP) and sensory action potential (SAP) will be analyzed according to the normative data in our laboratory. Studied nerves include bilateral median, ulnar, peroneal, tibial, and sural nerves. Abnormal result on NCS is defined as having abnormalities of 1 or more nerves with reduced amplitude, prolonged distal latency, or slowed nerve conduction velocity. Neurophysiologic criteria of sensorimotor polyneuropathy are defined as having symmetrical abnormalities in motor and sensory nerves (Dyck et al., 1985).

Tests of the autonomic nervous system. Sudomotor function will be examined using the sympathetic skin response (SSR) (Ravits, 1997). Results of SSR in the palm and sole will be interpreted as present or absent, but will not be evaluated quantitatively because of variations in the latencies and amplitudes of SSR. Parasympathetic function will be evaluated using the beat-to-beat heart rate variation [RR interval variability (RRIV)] at rest and during deep breathing (Ravits, 1997). Each test will be performed three times, and the mean value will be compared with that for the age-matched controls in our laboratory. Medication that interferes with sympathetic or parasympathetic functions will not be administered before or during these tests.

Statistical analysis. Numerical variables following Gaussian distribution will be compared using t-test and expressed as the mean  SD; for those variables not following Gaussian distribution, data will be expressed as the median (range) and will be analyzed with non-parametric Mann-Whitney U test. Results are considered significant if p < 0.05.

Patients with evidences of CNS disorders will be excluded first. Furthermore, those with attributable etiologies for neuropathy, such as diabetes, uremia, autoimmune disorders, or neoplasm will be excluded, too. The rest alcoholic patients will be separated as 2 groups: alcoholic patients with normal thiamine level (ATN) and alcoholic patients with thiamine deficiency (ATD). In the ATN group, patients will be further subgrouped as alcoholic patients without clinical evidence of neuropathy, alcoholic patients with sensory symptoms (especially burning lightning pains and painful paresthesia), and alcoholic patients with sensory and motor symptoms.

The first point to address in our study is to evaluate the prevalence of peripheral neuropathy in chronic alcoholic patients with emphasis on small-fiber involvement. Since early detection of neural degeneration is important, the sensitivity of punch skin biopsy, QST, NCS, and SSR and RRIV tests will be compared. The correlations between END and psychophysic and electrodiagnostic parameters will be discussed.

Second, we will elucidate the clinical significance of END reduction in alcoholic patients. END will be correlated with clinical manifestations and neurological deficits. Small-fiber sensory symptoms and signs will be correlated with END, and autonomic symptoms and signs will be correlated with the presence of sweat gland denervation. The degrees of END reduction in the 3 groups of ATN patients and control subjects will be compared. Since other systemic disease, especially diabetes, also causes small-fiber degeneration, we will examine whether alcoholic patients with diabetes have further cutaneous denervation.

Finally, the role of ethanol and thiamine in alcoholic neuropathy will be explored. The reduction of END will be correlated with thiamine status, lifetime ethanol dose, ethanol level, and other laboratory parameters. If END correlates with ethanol consumption, it will support the conclusion that alcoholic neuropathy is caused by direct toxic effect of ethanol or its metabolites. Since previous report documented the large-fiber-predominant axonal loss in sural nerve specimens in patients with pure-form of thiamine-deficiency neuropathy (Koike et al., 2003), we wonder if thiamine level influences small-fiber degeneration, i.e., reduction of END. The degrees of END reduction between alcoholic patients with ATD and those with ATN will be compared. These will further clarify the role of thiamine in alcoholic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria include daily uptake of at least 100 g ethanol for more than 3 years prior to the onset of neuropathic symptoms

Exclusion Criteria:

- Conditions known to be associated with peripheral neuropathy, such as diabetes, uremia, alcoholism, and the administration of potentially neurotoxic agents, such as alkylating agents, methotrexate, cyclosporine, and antibiotics, were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Tsung Tseng, MD, Study Director — 21,Nan-Yas S. Road. Sec 2 Pan-Chiao, Taipei, Taiwan; Sung-Tsang Hsieh, MD, PhD, Study Director — Department of Anatomy and Cell Biology, National Taiwan University College of Medicine, 1 Jen-Ai Road., Taipei 100, Taiwan
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taipei, Taiwan